CLINICAL TRIAL: NCT06273618
Title: iLookOut for Child Abuse: PA Microlearning to Improve Knowledge Retention
Brief Title: iLookOut Micro-learning to Improve Knowledge Retention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin H. Levi, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: iLO-ML-23396
Record Dates: First submitted 2023-12-30; First posted 2024-02-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Knowledge; Attitudes; Practice
Keywords: child maltreatment; suspicion of abuse; knowledge; attitudes; behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Early Childhood Professionals (ECPs) will be randomized to 1 of 4 groups, which will differ in terms of when they receive access to Micro-Learning. Non-ECPs will constitute a separate group, which will receive access to Micro-Learning immediately upon completing the Core Training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Immediate (Active Comparator): ECP participants who receive access to the Micro-Learning intervention immediately upon completing the Core Training.
  Interventions: Other: Micro-Learning
- 3-month (Active Comparator): ECP participants who receive access to the Micro-Learning intervention 3 months after upon completing the Core Training.
  Interventions: Other: Micro-Learning
- 6-month (Active Comparator): ECP participants who receive access to the Micro-Learning intervention 6 months after upon completing the Core Training.
  Interventions: Other: Micro-Learning
- 9-month (Active Comparator): ECP participants who receive access to the Micro-Learning intervention 9 months after upon completing the Core Training.
  Interventions: Other: Micro-Learning
- Non-ECPs (Active Comparator): Non-ECP participants
  Interventions: Other: Micro-Learning

INTERVENTIONS:
Other: Micro-Learning — Micro-Learning involves a series of 5-10 minute interactive, gamified learning exercises delivered to smart-phones (or computers) to reinforce and augment knowledge and promote attitudes and behavior to promote children's wellbeing.

SUMMARY:
This project investigates whether a multi-faceted strategy involving iLookOut's evidence-based Core Training plus an innovative follow-up Micro-Learning can promote knowledge retention and change behavior among early childhood professionals (ECPs) with regard to child abuse and its reporting. Additionally, this study will evaluate if non-ECPs experience similar improvements and retention of knowledge and changes in behavior as do ECPs.

DETAILED DESCRIPTION:
The primary purpose of this study is to understand the optimal timing to administer iLookOut Micro-Learning to boost ECPs waning knowledge and preparedness to protect children from abuse. Additionally, this study will conduct a randomized controlled trial to examine how interactive, gamified micro-learning promotes knowledge retention and fosters behavior change with regard to child abuse and its reporting, and to establish that implementation of this intervention is feasible.

All components of the learning module being studied are online, and will be accessed by participants through a secure website.

Once they complete the Core Training, participants who identify as ECPs will receive an email indicating which randomization arm they are in (regarding access to the advanced training) - immediate, 3 months, 6 months, or 9 months. Non-ECPs will be able to complete the advanced training as soon as they complete the Core Training. All non-ECPs will be used as a comparison group to determine if the iLookOut trainings are effective for improving and retaining knowledge, and changing behavior among Non-ECPs compared to the ECP participants.

Separate mixed-effects linear regression model will be applied to assess (1) the knowledge decay effect based on the data collected at different time-points and (2) the behavior change between the various time-points and how it is correlated to the knowledge score, after controlling for participants' baseline characteristics and work setting. In addition, the regression model will adjust effects for allocation blocks and the factors for stratification in the analysis to reduce group variability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Younger than 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge about child maltreatment and its reporting as assessed by validated iLookOut knowledge test | 3 months
  Validated knowledge test regarding child maltreatment and its reporting
Change in behavior regarding child maltreatment and its reporting as measured by self-report questionnaire | 3 months
  Self-report questionnaire of behavior regarding child maltreatment and its reporting

SECONDARY OUTCOMES:
Comparison of early childhood professionals vs. non-early childhood professionals | 6 months
  Comparison knowledge and behavioral outcomes for early childhood professionals vs. non-early childhood professionals

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will make available de-identified study data for the primary and secondary outcomes for authorized research projects upon request.